CLINICAL TRIAL: NCT02290795
Title: Vitreopapillary Traction and Optic Disc Morphology in Healthy Subjects, Vitreomacular Traction Patients and Glaucoma Patients
Brief Title: Vitreopapillary Interface and Optic Disc Morphology
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: VPI study
Record Dates: First submitted 2014-10-29; First posted 2014-11-14 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Posterior Vitreous Detachment; Vitreomacular Traction; Glaucoma; Vitreopapillary Traction
Keywords: Vitreopapillary traction
MeSH Terms: conditions — Vitreous Detachment; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- healthy subjects: Healthy subjects (not diagnosed with any eye disease affecting the vitreous or optic nerve head).
  Interventions: Other: OCT imaging/HRT imaging
- Glaucoma patients: Glaucoma patients visiting the glaucoma consultation.
  Interventions: Other: OCT imaging/HRT imaging
- Patients scheduled for trabeculectomy: Glaucoma patients scheduled for filtering surgery (=trabeculectomy)
  Interventions: Other: OCT imaging/HRT imaging
- Vitreomacular traction patients: Patients with symptomative vitreomacular adhesion scheduled for treatment with Ocriplasmin
  Interventions: Other: OCT imaging/HRT imaging

INTERVENTIONS:
Other: OCT imaging/HRT imaging — Standard follow up protocol with Optical coherence Tomography (OCT) imaging and Heidelberg Retinal Tomograph (HRT) imaging for glaucoma patients and patients scheduled for Ocriplasmin treatment In case of healthy controls the same investigations will be performed.

SUMMARY:
The vitreous fills the posterior chamber of the eye and is firmly attached, at the posterior pole, to the macula and the optic nerve head (ONH). With formation of a stepwise posterior vitreous detachment (PVD) exerted tractional forces could influence retinal functioning. Especially in patients with glaucoma the influence of vitreous traction to the ONH could mask progression, interfere with current imaging techniques and even be a cause of ONH hemorrhages. Therefore the aim of this study is to investigate whether vitreopapillary traction has a significant effect on diagnosis and follow up of glaucoma patients.

DETAILED DESCRIPTION:
The vitreous body fills the posterior chamber of the eye and consists mainly of water. It is kept organized into a gel like structure by numerous collagen fibrils and makes contact with the surrounding retina. This interplay known as the vitreo-retinal interface of the human eye is a complex organization of bridging molecules anchoring the vitreous to the internal limiting membrane. With ageing, the vitreous gel undergoes liquefaction accompanied by progressive weakening of the adhesions at the vitreo-retinal interface resulting in a stepwise process of adhesion release. Since the most firm attachments in the posterior pole are situated at the macular and papillary region, tractional forces exerted during vitreous separation could influence retinal functioning.

Up until now researchers have been looking primarily at the influence of vitreous traction to the macular region of the nerve fiber layer.This research has led to the insight that vitreo-macular traction can result in macular hole formation, and that patients with this condition may benefit from vitreolysis induced by surgery (vitrectomy) or intravitreal injection of ocriplasmin.

More recent reports have focused on the influence of the vitreous on the morphology of the optic disc, showing that VPT altered optic disc architecture, increased average and temporal retinal nerve fiber layer thickness and was associated with more pronounced visual field defects. This could be important as very sensitive scans and diagnostic algorithms were developed for staging and follow up of glaucoma patients' optic nerve head, which could be influenced by the patients' vitreopapillar interface. As the status of this interface changes over time, this could lead to confusion and misinterpretation of the optic disc diagnostic scans.

Besides the diagnostic challenges induced by the vitreopapillar interaction, this interface may also be of pathogenetic relevance in glaucoma. Indeed, the optic disc represents the collection of all ganglion cell axons, and glaucoma is caused by a degeneration of ganglion cells. Some authors have already suggested that vitreopapillary traction (VPT) could play a role in the pathogenesis of optic nerve head hemorrhages, which are regarded as an important risk factor for glaucoma progression. Moreover, one could hypothesize that VPT can cause stress to the ganglion cell axons and therefore contribute more directly to ganglion cell degeneration.

Accordingly, this study aims at investigating the effect of VPT on the ultra-structural level of the optic disc. A possible structure-function relation will be investigated with the help of central visual field tests and focal retinal nerve fiber layer thickness assessment. With increasing knowledge and imaging of VPT, possibly a VPT-staging algorithm can be developed and VPT risk factors defined. Finally, this project may have a therapeutic impact, since it will shed light on the question whether (surgically or chemically) induced vitreolysis might be beneficial in some glaucoma patients with VPT.

ELIGIBILITY:
Inclusion Criteria:

* willingness to sign informed consent, aged over 18y, glaucoma/trabeculectomy scheduled/Ocriplasmin scheduled/healthy

Exclusion Criteria:

* medical history of vitrectomy/diabetes/Retinal Vessel Occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients visiting either the glaucoma consultation or the vitreo-retinal disease consultation (depending on study group recruitment). Healthy controls will be recruited from subjects accompanying these patients.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of VPT in glaucoma patients | From inclusion up to 17 months
  Percentage of patients diagnosed with glaucoma who have Vitreopapillary traction.
Change in VPT following trabeculectomy | From inclusion up to 17 months with an average follow up of 8 weeks per subject
  To investigate whether the sudden decrease in intraocular pressure following trabeculectomy has a significant effect on ONH morphology (mean retinal nerve fiber layer (mRNFL) thickness, cup volume, rim thickness, cup/disc ratio) caused by change in VPT. Patients scheduled for trabeculectomy will have a baseline visit up until 8 weeks before the surgery and 4 post operative visits (day 1, week 1, 2 and 4)
Change in VPT following ocriplasmin | From inclusion up to 17 months with an average follow up of 8 weeks per subject
  To investigate whether the use of Ocriplasmin has a significant effect on ONH morphology (mRNFL thickness, cup volume, rim thickness, cup/disc ratio) caused by change in VPT. Patients scheduled for Ocriplasmin treatment will have a baseline visit 1 week before the surgery and 2 post operative visits (day 1, week 4)

SECONDARY OUTCOMES:
Proportion of patients with VPT that present with optic nerve head hemorrhage | From inclusion up to 17 months
  To investigate whether patients with VPT have significantly more chance of ONH hemorrhages than subjects without VPT. Cross-sectional analysis so 1 visit per patient between 11/2014 and 4/2016.
Proportion of patients with focal visual field defect that have corresponding focal VPT | From inclusion up to 17 months
  To investigate whether a firm vitreous attachment and traction to a certain part of the ONH (focal rim thickness, focal RNFL thickness) could play a role in the formation of anatomically linked visual field defects. Cross-sectional analysis so 1 visit per patient between 11/2014 and 4/2016. Part two of the analysis on patients scheduled for trabeculectomy who will have a baseline visit up until 8 weeks before the surgery and 4 post operative visits (day 1, week 1, 2 and 4)

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD PhD, Principal Investigator — Dpt. Ophthalmology, University Hospitals Leuven, Belgium
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Kim YW, Jeoung JW, Yu HG. Vitreopapillary traction in eyes with idiopathic epiretinal membrane: a spectral-domain optical coherence tomography study. Ophthalmology. 2014 Oct;121(10):1976-82. doi: 10.1016/j.ophtha.2014.04.011. Epub 2014 May 29. PMID 24880904
- [Background] Wisotsky BJ, Magat-Gordon CB, Puklin JE. Vitreopapillary traction as a cause of elevated optic nerve head. Am J Ophthalmol. 1998 Jul;126(1):137-9. doi: 10.1016/s0002-9394(98)00080-4. PMID 9683164
- [Background] Hwang YH, Kim YY. Peripapillary retinal nerve fiber layer thickening associated with vitreopapillary traction. Semin Ophthalmol. 2015 Mar;30(2):136-8. doi: 10.3109/08820538.2013.833257. Epub 2013 Oct 30. PMID 24171792
- [Derived] Willekens K, Abegao Pinto L, Lemmens S, Bataillie S, Somers A, Vandewalle E, Stalmans P, Stalmans I. The vitreopapillary interface in healthy and glaucoma: posterior vitreous detachment in the vitreopapillary interface study. Acta Ophthalmol. 2018 Sep;96(6):573-581. doi: 10.1111/aos.13818. Epub 2018 Oct 2. PMID 30280516